CLINICAL TRIAL: NCT06893523
Title: Evaluation of the Effect of Concentrated Growth Factor (CGF) on Postoperative Edema in Bilateral Impacted Third Molar Surgery: A Randomized Controlled Clinical Study
Brief Title: Effect of CGF on Postoperative Edema in Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mert Zeytinoğlu, Assoc. Prof. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGE-DHF-MZ-001
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Oral Complication
Keywords: Edema; Third molar
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGF (Experimental): Participants received CGF after the operation on one side
  Interventions: Other: Concentrated Growth Factor; Other: Non-CGF
- non-CGF (No Intervention): The other extraction socket is left empty

INTERVENTIONS:
Other: Concentrated Growth Factor — Bilaterally impacted third molar of the patients areremoved surgically and concentrated growth factor isplaced in one of the extraction sockets.
  Arms: CGF
Other: Non-CGF — The other extraction socket is left empty for control purposes.
  Arms: CGF

SUMMARY:
The purpose of this study is to evaluate the effects of concentrated growth factor (CGF) on edema after bilateral impacted third molar surgery and to determine its contribution to the healing process.

The main question it aims to answer is:

Is CGF effective on reducing the edema in impacted third molar surgery? Researchers compare the edema amount on the CGF-applied and CGF free sides after impacted third molar surgery. The edema measurements are performed on the second and seventh days.

DETAILED DESCRIPTION:
It has been observed that the treatment of impacted tooth extraction, which is the most commonly performed interventional procedure in oral and maxillofacial surgery clinics and affects the patient's comfort and daily life after the operation, has been investigated in many ways and new ideas are constantly emerging. Wound healing is a process controlled by many intracellular and extracellular mechanisms. In recent years, many studies have been conducted to make this process faster and more successful, and it has been observed that the use of platelet products in this area has yielded extremely successful results. Concentrated Growth Factor (CGF), which has gained an important place in regenerative medicine in recent years, has attracted attention due to its potential to minimize postoperative complications.

This randomized clinical trial was conducted at the Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Ege University.

Forty-nine patients, regardless of gender, with bilateral, symmetrical, bone-retained (vertical, mesioangular, horizontal) impacted third molar in the mandible and without any systemic disease are included in the study. Before the impacted third molar surgery, detailed medical and dental history are taken from the patients.

The patients are informed in detail about the drugs to be used in the study, the applied method, the duration and purpose of the study.

In order to obtain the data required for statistical analysis of the amount of edema on the sides where CGF is used and not used after the operation, edema measurements are made at three points on the patients before the operation, on the 2nd and 7th days after the operation.

These measurements are made between the external canthus-angulus mandible, tragus-commissura and tragus-pogonium.

Wilcoxon Signed Ranks test is used to compare the means of two dependent samples and to determine the significance of the difference between them.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral, symmetrical, bone-retained (vertical, mesioangular, horizontal) impacted wisdom teeth in the mandible, regardless of gender
* Patients without any systemic disease
* Patients who have been informed about the duration, purpose and requirements of the study and who have signed the informed consent form voluntarily.-

Exclusion Criteria:

* Having a disease affecting general health that requires the application of prophylactic antimicrobial agents
* Having a systemic viral, fungal or bacterial infection
* Patients with acute or chronic maxillary sinusitis
* Suspected or diagnosed pregnancy and nursing mothers
* Patients with heart and vascular diseases
* Patients with liver disease, haematological disease and neoplastic disease
* Patients who have recently received anti-inflammatory therapy
* Patients with chronic medication use (antihistamines, NSAIDs, steroids and antidepressants)
* Patients predisposed to psychotic or psychopathic tendencies
* Patients with rheumatic diseases, blood diseases, diabetes mellitus
* Patients at cardiological risk of infective endocarditis
* Patients under antibiotic pressure

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Postoperative edema amounts on CGF-applied and CGF free sides in bilateral impacted third molar surgery | Before operation to the end of the operation at seven days
  Edema measurements are made at three points on the patients before the operation, on the 2nd and 7th days after the operation. These measurements are made between the external canthus-angulus mandible, tragus-commissura and tragus-pogonium. In order to ensure standardization, all measurements are made by the same physician with the patient's head position in the same direction.

CONTACTS AND LOCATIONS:
Overall Officials: Mert Zeytinoglu, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Dentistry, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No